CLINICAL TRIAL: NCT04487223
Title: Characterization of Novel Lipoprotein Properties Associated With an Increased Risk to Develop Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Rom Keshet, Principal Investigator, Sheba Medical Center
Other Study IDs: 6500-19-SMC
Record Dates: First submitted 2020-07-07; First posted 2020-07-27 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives of Medical Research:

Separation of LDL and HDL from blood samples of patients with high LDL and / or low HDL who have developed atherosclerotic disease with similar patients who have no evidence of atherosclerosis.

Lipidomics and proteomics will examine whether there is a difference in lipid and protein composition and lipoprotein composition. If there are any changes in expression level or the composition of proteins or metabolites that make up lipoproteins, the investigator will try to figure out the mechanism responsible for these changes and their role in the metabolic process. the investigator will seek therapeutic measures through which these mechanisms can be inhibited and thus inhibit the development of sclerosis or even retraction.

DETAILED DESCRIPTION:
Participants:

Participants who are found suitable during their visit to the Lipid Institute Clinic or during hospitalization at the Sheba Medical Center will receive an explanation of the study, will be asked to sign a consent form.

A medical history will be taken, the participant will be asked to fill out a nutrition questionnaire (FFQ) and a 5 cc blood sample will be taken from each patient

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with LDL levels less than 130 mg / dl without evidence of atherosclerosis or wall thickening of the carotid artery according to an ultrasound imaging of the carotid artery at the Lipid Institute and unknown for atherosclerosis or cardiovascular disease in the background.
* Participants with LDL levels above 160 mg / dl, with no evidence of atherosclerosis or wall thickening of the carotid artery according to an ultrasound - IMT of the carotid arteries performed at the Lipid Institute and unknown for atherosclerosis or cardiovascular disease in the background.
* Participants with LDL levels above 160 mg / dl, where evidence of atherosclerosis or wall thickening of the arteries can be found by ultrasound imaging of the carotid artery that is performed at the Lipid Institute or known for atherosclerosis or cardiovascular disease in the background.

Exclusion Criteria:

* Patients with triglyceride values above 300 mg%, HDL lower than 30 mg%, APOB greater than 150 mg% or LPa higher than 70 mg% will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at the Sheba Medical Center's Lipid Institute, participants will be the Lipid Institute's patients Number of participants: 20 patients with hypercholesterolemia and sclerosis, 20 patients with hypercholesterolemia without evidence of sclerosis, 20 healthy participants as a control group.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-04-27 (Estimated); Study Completion 2022-04-27 (Estimated)

PRIMARY OUTCOMES:
Characterization of novel lipoprotein properties associated with an increased risk to develop atherosclerosis | 1 year
  Lipoproteins would be analyzed by lipidomic and proteomic profiling using chromatography and mass-spectrometry. Concentrations of specific lipids and proteins will be quantified as micrograms per deciliter or as area under the curve. We will look for significant differences in these values between the different study groups using updated software tools specifically designed for mass spectrometry data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Lipid center, Tel Litwinsky, Israel